CLINICAL TRIAL: NCT00996359
Title: Partially HLA-Matched Irradiated Allogeneic Cellular Therapy After Reduced Intensity Total Body Irradiation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020901; P30CA072720 (NIH); CDR0000656757 (Other: NIH); IRB# 0220090213
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; adult acute myeloid leukemia in remission; recurrent adult acute lymphoblastic leukemia; adult acute lymphoblastic leukemia in remission; relapsing chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; chronic myelomonocytic leukemia; recurrent adult diffuse large cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; adult nasal type extranodal NK/T-cell lymphoma; peripheral T-cell lymphoma; hepatosplenic T-cell lymphoma; anaplastic large cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; childhood diffuse large cell lymphoma; recurrent childhood large cell lymphoma; Burkitt lymphoma; childhood immunoblastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood anaplastic large cell lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood small noncleaved cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Blast Crisis; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelomonocytic, Chronic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Lymphoma, T-Cell, Peripheral; Lymphoma, Large-Cell, Anaplastic; Hodgkin Disease; Dendritic Cell Sarcoma, Interdigitating; Immunoblastic Lymphadenopathy | interventions — Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irradiated allogeneic lymphocytes after Total Body Irradiation (Experimental)
  Interventions: Biological: Irradiated haploidentical allogeneic lymphocytes; Radiation: total-body irradiation

INTERVENTIONS:
Biological: Irradiated haploidentical allogeneic lymphocytes — Partially HLA-matched irradiated donor lymphocytes will be infused after total body irradiation.
Radiation: total-body irradiation — 100 cGy TBI

SUMMARY:
RATIONALE: Giving low-dose total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect).

PURPOSE: This phase I trial is studying the side effects of donor stem cell transplant after total-body irradiation and to see how well it works in treating patients with relapsed or refractory hematologic cancer or acute myeloid leukemia or acute lymphocytic leukemia in complete remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the toxicity of irradiated haploidentical allogeneic cellular therapy after low-dose total-body irradiation and no pharmacologic graft-vs-host disease prophylaxis in patients with relapsed or refractory hematologic malignancies or patients with acute myeloid leukemia (AML) or acute lymphoblastic leukemia in second or greater complete remission (CR2).

Secondary

* To evaluate immunologic parameters before and after haploidentical therapy.
* To demonstrate host anti-leukemia T-cells in a subset of patients with AML who are HLA-A2-positive.
* To observe any evidence of antitumor activity within the confines of this pilot study and/or assess the duration of remission in those patients who enter the study in CR2.

OUTLINE: Patients undergo low-dose total-body irradiation and infusion of irradiated donor cells on day 0. Patients also receive filgrastim subcutaneously (SC) daily or pegfilgrastim SC every 14 days starting on day 1.

Patients in complete remission (CR) or with persistent disease undergo irradiated donor lymphocyte infusion (DLI) at 8 weeks. Repeat irradiated DLI is administered if patients remain in CR or achieve stable or responding disease after the second infusion (if confirmed by histologic assessment) or third infusion (if confirmed by radiographic assessment). DLI repeats every 8 weeks pending disease and clinical status up to a total of 6 infusions over a 12-month period.

Blood samples are collected at baseline, upon recovery of counts, and then monthly thereafter for immunologic studies.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients over 18 years old must meet the following criteria:

  * Histologically confirmed hematologic malignancy and not a candidate for a standard allogeneic transplantation
  * High-risk disease, including:

    * Refractory/relapsed acute myeloid leukemia (AML) or AML in second or greater completion remission (CR2)
    * Relapsed or refractory acute lymphoblastic leukemia (ALL) or ALL in CR2
    * Tyrosine kinase inhibitor-resistant chronic myelogenous leukemia in chronic, accelerated, or blast crisis
    * Fludarabine-resistant chronic lymphocytic leukemia
    * High-risk myelodysplastic syndrome (MDS) (i.e., MDS with a score ≥ 1.5 by the International Scoring System)
    * Chronic myelomonocytic leukemia
    * Relapsed diffuse large cell non-Hodgkin lymphoma (NHL) with measurable disease after (or not eligible for) high-dose chemotherapy/autologous hematopoietic stem cell (HSC) rescue or allogeneic hematopoietic stem cell transplantation (HSCT)
    * Relapsed follicular NHL, mantle cell lymphoma, or low-grade histology NHL with measurable disease after (or not eligible for) high-dose chemotherapy/autologous HSC rescue or allogeneic HSCT
    * Relapsed or refractory high-grade/aggressive NHL (Burkitt lymphoma, lymphoblastic lymphoma, T-cell lymphoma, NK-like lymphoma) with measurable disease after (or not eligible for) high-dose chemotherapy/autologous HSC rescue or allogeneic HSCT
    * Hodgkin lymphoma with measurable disease after (or not eligible for) high-dose chemotherapy/autologous HSC rescue or allogeneic HSCT
    * Relapsed or refractory multiple myeloma after (or not eligible for) high-dose chemotherapy/autologous HSC rescue and following salvage therapy with thalidomide, lenalidomide, bortezomib or other FDA-approved multiple myeloma salvage therapies
* Patients 13-17 years old must meet the following criteria:

  * Histologically confirmed hematologic malignancy and not a candidate for a standard allogeneic transplantation
  * High-risk disease, including:

    * Refractory/relapsed AML or AML in CR2
    * Relapsed or refractory ALL or ALL in CR2
    * Relapsed diffuse large cell NHL with measurable disease after (or not eligible for) high-dose chemotherapy/autologous HSC rescue or allogeneic HSCT
    * Relapsed follicular NHL, mantle cell lymphoma (or low-grade histology NHL) with measurable disease after (or not eligible for) high-dose chemotherapy/autologous HSC rescue or allogeneic HSCT
    * Relapsed or refractory high-grade/aggressive NHL (Burkitt lymphoma, lymphoblastic lymphoma, T-cell lymphoma, NK-like lymphoma) with measurable disease after (or not eligible for) high-dose chemotherapy/autologous HSC rescue or allogeneic HSCT
    * Hodgkin lymphoma with measurable disease after (or not eligible for) high-dose chemotherapy/autologous HSC rescue or allogeneic HSCT
* Eligible for haploidentical irradiated cellular therapy
* No known active brain metastases or malignant meningitis
* Available partially (≥ 3/6 class I antigen) HLA-matched (by serology) related donor NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2
* Karnofsky PS 60-100% (for patients > 16 years) or Lansky PS 60-100% (for patients ≤ 16 years)

  * Patients who are unable to walk because of paralysis but who are up in a wheelchair will be considered ambulatory for the purpose of assessing PS
* Patients ≥ 18 years:

  * Total bilirubin < 1.5 times upper limit of normal (ULN) (unless attributable to Gilbert disease)
  * DLCO/alveolar volume > 50%
  * Serum creatinine < 2.0 mg/dL
* Patients 13-17 years:

  * Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age/gender as follows:

    * 13 to < 16 years: 1.5 mg/dL (male) or 1.4 mg/dL (female)
    * ≥ 16 years: 1.7 mg/dL (male) or 1.4 mg/dL (female)
  * AST/ALT ≤ 2.5 times ULN for age
  * Total bilirubin < 2.0 mg/dL (unless attributable to Gilbert syndrome)
  * Shortening fraction ≥ 27% by ECHO or ejection fraction ≥ 50% by radionuclide angiogram
  * FEV_1, forced vital capacity, and DLCO corrected for hemoglobin ≥ 60% by pulmonary function tests (PFTs)

    * Children unable to cooperate for PFTs must meet the following criteria:

      * No evidence of dyspnea at rest
      * No exercise intolerance
      * No requirement for supplemental oxygen therapy
  * Any other organ dysfunction thought to be secondary to disease will be considered separately and the patient will be eligible at the physician's discretion
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for 24 weeks after study treatment
* No known HIV positivity
* No history of current or prior medical problems that, in the investigator's opinion, would prevent administration of study treatment or assessment of response due to excess toxicity
* No active uncontrolled infections or other medical, psychological, or social conditions that might increase the likelihood of patient adverse effects or poor outcomes

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No corticosteroids within 2 weeks before receiving irradiated donor lymphocyte infusion
* No medications that might increase the likelihood of patient adverse effects or poor outcomes

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Toxicity | 3 years

SECONDARY OUTCOMES:
Immunologic parameters before and after haploidentical therapy | 3 years
Anti-tumor activity and/or duration of remission in those patients who enter the study in second complete remission or greater | 3 years
Treatment-related mortality | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States